CLINICAL TRIAL: NCT00302796
Title: Antibiotic Treatment to Patients With Low Back Pain Associated With Modic Changes Following Disc Herniation. A Randomized Clinical Controlled Trial
Brief Title: Antibiotic Treatment to Patients With Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Back Research Center, Denmark (Other)
Responsible Party: Hanne Albert, The Back Research Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-005500-17
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-07

CONDITIONS: Back Pain
Keywords: Low Back Pain,
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A, Antibiotic (Experimental): 1 antibiotic tablet 45 patients Group
  Interventions: Drug: Bioclavid
- Group B: 1 placebo (Placebo Comparator): 1 placebo tablet
  Interventions: Drug: Placebo
- Group C: Antibiotics (Experimental): 2 antibiotic tablets 45 patients
  Interventions: Drug: Bioclavid
- Group D, Placebo (Placebo Comparator): 2 placebo tablets 36 patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bioclavid — 500 + 125 mg times 3 or 6
  Arms: Group A, Antibiotic; Group C: Antibiotics
Drug: Placebo
  Arms: Group B: 1 placebo; Group D, Placebo

SUMMARY:
A large proportion of patients with Low Back Pain (LBP) (80 %) are classified as "non-specific", due to the lack of a patho-anatomical diagnosis. This term is not satisfactory, since it implies uncertainty for both the patient and the clinician. Modic changes have recently been identified as a pain giving patho-anatomical diagnosis for a considerable percentage (20-30 %) of LBP patients. The causes of these Modic changes have not been determined conclusively but bacterial infection is among the plausible causes for those following a disc herniation.

Purpose The aim of this study is to assess the clinical effect of antibiotic treatment compared to placebo, in patients with LBP and Modic changes following a lumbar herniated disc.

Design A double blind prospective clinically controlled trial. Patients will be randomized by a blinded observer to either Group A: 1 antibiotic tablet 45 patients Group B: 1 placebo tablet 36 patients Group C: 2 antibiotic tablets 45 patients Group D: 2 placebo tablets 36 patients

The patients will take the drug three times a day for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Previous lumbar herniated disc confirmed by MRI
* Time since lumbar disc herniation more than 6 months less than 2 years
* LBP in the area of L1 to L5, with an added Low Back Pain Rating Scale of 6 or more
* The present MRI shows Modic changes
* Positive Springing test (SPT) at the level of Modic changes

Exclusion Criteria:

* Allergy against antibiotics
* The Beck Depression Inventory >7,
* Pregnancy
* Breast feeding
* All Kidney diseases
* Pending workers litigation or pension
* Danish as second language
* Fertile women who do not user safe anti conseption
* Reduced liver functions
* Reduced liver function due to previous treatment wiht amoxicillin/clavulanasid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Low Back Pain Roland Morris Questionaire | One year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hanne B Albert, Ph.D, Principal Investigator — The Back Research Center, University of Southern Denmark
Locations (1):
- The Back Research Center, Ringe, Denmark